CLINICAL TRIAL: NCT00452712
Title: Orthostatic Hypotension in Children With Acute Febrile Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 156/06
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Fever; Orthostatic Hypotension
Keywords: orthostatism; fever
MeSH Terms: conditions — Fever; Hypotension, Orthostatic | interventions — Supine Position; RE1-silencing transcription factor; Standing Position

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: All subjects will have their blood pressure measured in supine position (after 5 minute of rest) and after 3 minute of standing.

SUMMARY:
Objective:to determent if children suffering from acute febrile illness has higher rate of orthostatic hypotension compared with children with no febrile illness. Design: a prospective cohort study. Subjects: children aged 4-18 year with fever (temperature > 38.) for up to 48 hours, presenting to the pediatric emergency department. Interventions: All subjects will have their blood pressure measured in supine position (after 5 minute of rest) and after 3 minute of standing.

DETAILED DESCRIPTION:
Orthosatic hypotension describes a condition in which the autonomic nervous system fails to maintain a stable blood pressure in the face of postural change. Children presenting to the pediatric ED with fever often describe symptom like syncope, lightheadedness, dizziness, pallor, fatigue and weakness. These symptom may result from orthostatism related to acute febrile illness. We assume that fever may be associated with autonomic changes (e.g. vasodilatation) that can cause orthostatism. Objective:

to determent if children suffering from acute febrile illness has higher rate of orthostatic hypotension compared with children with no febrile illness. Design: a prospective cohort study. Subjects: children aged 4-18 year with fever (temperature > 38.) for up to 48 hours, presenting to the pediatric emergency department. Interventions: All subjects will have their blood pressure measured in supine position (after 5 minute of rest) and after 3 minute of standing. Data analysis: The proportion of children with orthostatic hypotension in febrile and non febrile patients will be compared using χ2 test. The changes in blood pressure in both groups will be compared using the Student t test.

Assumption: We assumed that the incidence of orthostatism is higher among children with fever, because fever can cause orthostatism. Significance: Orthostatism can cause syncope which is a potentially dangerous symptom (e.g. head trauma). Syncope accounts for 1-3% of hospital admissions in US. The incidence in youths is estimated at about 15%) Patients presenting to the ED with syncope may undergo numerous and expensive work up with low diagnostic yield. -understanding that fever itself can cause orthostatism and syncope may help us with precaution and diagnosis.

Key word: orthostatism, fever children, emergency medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4-18 year of age.
* Oral temperature > 38.0
* Duration of fever 6-48 hours

Exclusion Criteria:

* Treatment with medications that may cause orthostatism.
* Vomiting or/and diarrhea (more than twice/day).
* Suspected CNS infection.
* Chronic diseases
* Unable to give an informed consent

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kozer, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel